CLINICAL TRIAL: NCT00611442
Title: Single Dose Lubiprostone Along With Split-dose PEG Solution Without Dietary Restrictions for Bowel Cleansing Prior to Colonoscopy, a Randomized, Double-blind, Placebo Controlled Trial
Brief Title: Split Dose Golytely With Amitiza Pretreatment Versus Split Dose Golytely Plus Placebo in Outpatient Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Joel Z. Stengel, Gastroenterology Fellow, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.2007.188; IND 78254
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Results first posted 2012-11-01 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Bowel Preparation for Colonoscopy
MeSH Terms: interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): split-dose PEG solution without dietary restrictions plus lubiprostone 24mcg gelcap pretreatment
  Interventions: Drug: lubiprostone
- 2 (Placebo Comparator): split-dose PEG solution without dietary restrictions plus placebo pretreatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lubiprostone — lubiprostone 24mcg gelcap, 1 gelcap taken at noon the day prior to the colonoscopy
  Other Names: amitiza
  Arms: 1
Drug: placebo — placebo gelcap, taken at noon the day prior to the colonoscopy
  Arms: 2

SUMMARY:
The primary outcomes of this procedure will be: 1. The cleanliness of the prep as measured by the Ottawa Scale (attachment a). Secondary outcomes will be: 1. Patient satisfaction with the prep measured by 5 point Likert scale (attachment b); 2. Procedure time; 3. The number and size of polyps detected on examination.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients referred to our clinic for Average or Increased Risk screening for Colorectal Cancer
* Ages will be from 18 years of age and older

Exclusion Criteria:

* Chronic kidney disease
* Previous diagnosis of congestive heart failure
* History of bowel obstruction
* History of solid organ transplant
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Z Stengel, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Harewood GC, Wiersema MJ, Melton LJ 3rd. A prospective, controlled assessment of factors influencing acceptance of screening colonoscopy. Am J Gastroenterol. 2002 Dec;97(12):3186-94. doi: 10.1111/j.1572-0241.2002.07129.x. PMID 12492209
- [Background] Tan JJ, Tjandra JJ. Which is the optimal bowel preparation for colonoscopy - a meta-analysis. Colorectal Dis. 2006 May;8(4):247-58. doi: 10.1111/j.1463-1318.2006.00970.x. PMID 16630226
- [Background] El Sayed AM, Kanafani ZA, Mourad FH, Soweid AM, Barada KA, Adorian CS, Nasreddine WA, Sharara AI. A randomized single-blind trial of whole versus split-dose polyethylene glycol-electrolyte solution for colonoscopy preparation. Gastrointest Endosc. 2003 Jul;58(1):36-40. doi: 10.1067/mge.2003.318. PMID 12838218
- [Background] Church JM. Effectiveness of polyethylene glycol antegrade gut lavage bowel preparation for colonoscopy--timing is the key! Dis Colon Rectum. 1998 Oct;41(10):1223-5. doi: 10.1007/BF02258217. PMID 9788383
- [Background] Lacy BE, Levy LC. Lubiprostone: a chloride channel activator. J Clin Gastroenterol. 2007 Apr;41(4):345-51. doi: 10.1097/01.mcg.0000225665.68920.df. PMID 17413599

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Gastroenterology Clinic, Brooke Army Medical Center, Fort Sam Houston, TX October 2007 to January 2008
Groups:
- Amitiza: split-dose PEG solution without dietary restrictions plus lubiprostone 24mcg gelcap pretreatment
- Placebo: split-dose PEG solution without dietary restrictions plus placebo pretreatment
Period: Overall Study
Arm/Group | Amitiza | Placebo
Started | 95 | 96
Completed | 94 | 94
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amitiza | Placebo | Total
Number analyzed (Participants) | 95 | 96 | 191
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 94 | 96 | 190
  >=65 years | 1 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 55.4 (5.2) | 55.9 (4.8) | 55.5 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 45 | 93
  Male | 47 | 51 | 98
Region of Enrollment [Number; unit: participants]
  United States | 95 | 96 | 191

OUTCOME MEASURES:

1. Primary Outcome: The Overall Cleanliness of the Prep as Measured by the Ottawa Scale
Description: Bowel cleansing was evaluated with the Ottawa bowel preparation scale by each endoscopist during the endoscopy. Neither the endoscopist nor the endoscopy nurse was aware of the bowel preparation used prior to the colonoscopy. The Ottawa bowel preparation scale is a validated tool and was used in this study to provide a reliable quality assessment of the bowel preparation used for colonoscopy. This validated scale rates each section of the colon, the right, the mid, and the rectosigmoid colon, on a 5-point scale (0-4), as well as a global 3-point rating for overall colonic fluid (0-2). The total score ranges from 0 to 14. An excellent preparation with little fluid would score 0-3, a good preparation 4-6, while scores higher than 7would indicate progressively worsening bowel preparations. A completely unprepared colon would score 11-14, depending on the amount of colonic fluid
Time Frame: measured upon completion of the colonoscopy, colonoscopies completed during the course of the study (approximately 4 month period)
Measure: Mean (Full Range); unit: Ottawa Score
Arm/Group | Amitiza | Placebo
Number analyzed (Participants) | 94 | 94
Ottawa Score | 4.8 [3 to 10] | 6.2 [3 to 12]

2. Secondary Outcome: Patient Satisfaction With the Prep Measured by 5 Point Likert Scale
Description: The participants completed a survey prior to the colonoscopy that graded their overall satisfaction with the bowel preparation. The subjects rated the survey questions on a 5-point Likert scale where 1 = severely distressing, 2=distressing, 3=bothersome, 4=mild, and 5=none.
Time Frame: measured after completion of the bowel preparation and prior to the colonoscopy, completed during the course of the study (approximately 4 month period)
Measure: Mean (Standard Deviation); unit: linkert scale (1-5)
Arm/Group | Amitiza | Placebo
Number analyzed (Participants) | 94 | 94
linkert scale (1-5) | 3.7 (1.0) | 3.2 (1.1)

3. Secondary Outcome: Procedure Time
Description: Procedure time refers to the total length of time required to complete the colonoscopy
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Amitiza | Placebo
Number analyzed (Participants) | 94 | 94
minutes | 17.8 (5.4) | 19.8 (6.2)

4. Secondary Outcome: The Number of Polyps Detected on Examination
Description: The number of colon polyps detected during the colonoscopy.
Time Frame: as for outcome 1
Measure: Number; unit: number of polyps
Arm/Group | Amitiza | Placebo
Number analyzed (Participants) | 94 | 94
number of polyps | 48 | 44

ADVERSE EVENTS:
Arm/Group | Amitiza | Placebo
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/94
Other Adverse Events (participants affected / at risk) | 0/94 | 0/94

LIMITATIONS AND CAVEATS:
This study may be limited by the recruitment of outpatients as the only study participants. The study results might have also been affected by limiting the indication for colonoscopy to colorectal cancer screening.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No